CLINICAL TRIAL: NCT01250834
Title: Effect of LY2189265 on the Pharmacokinetics of Atorvastatin in Healthy Subjects
Brief Title: LY2189265 and Atorvastatin Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11551; H9X-MC-GBCP (Other: Eli Lilly and Company); 2010-021657-39 (EudraCT Number)
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Atorvastatin; dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2189265 + Atorvastatin (Experimental): Period 1: Participants received a single 40-milligram (mg) oral dose of atorvastatin on Day 1, followed by a 7- to 10-day washout period between Period 1 and Period 2.
  Period 2: Participants received a single 1.5-mg subcutaneous dose of LY2189265 on Day 1, followed by a single 40-mg oral dose of atorvastatin on Day 3.
  Interventions: Drug: Atorvastatin; Biological: LY2189265

INTERVENTIONS:
Drug: Atorvastatin — Administered orally.
Biological: LY2189265 — Administered subcutaneously.

SUMMARY:
This study will assess if giving LY2189265 at the same time as atorvastatin affects how the body absorbs atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with female partners of child-bearing potential: Agree and whose partners agree to use two reliable methods of contraception from the time of the first dose until 3 months after the last dose of study drug, as determined by the investigator.
* Female subjects not of child-bearing potential (that is, are postmenopausal or permanently sterilized [for example, tubal occlusion, hysterectomy, bilateral salpingectomy]) will not be required to use contraception. Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) with follicle stimulating hormone (FSH) greater than or equal to 40 milliInternational Units per milliliter (mIU/mL).
* Female subjects who have undergone sterilization by tubal ligation: Agree to use a male or female condom used in conjunction with spermicidal gel, foam, cream, film or suppository from the time of screening until 3 months after the last dose of study drug. Such subjects must also test negative for pregnancy at the time of enrollment.
* Have a body mass index (BMI) between 18.5 and 30.0 kilograms per square meter (kg/m^2), inclusive.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow frequent blood sampling.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow the study restrictions

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 90 days from a clinical trial involving an investigational drug or device or off-label use of a drug or device or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies or intolerance to atorvastatin.
* Have known allergies to glucagon-like peptide-1 (GLP-1)-related compounds including LY2189265.
* Are persons who have previously completed or withdrawn from this study, or have taken part in any other study investigating LY2189265 or GLP-1-related compounds or incretin mimetics within the last 3 months.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure (after at least 5 minutes sitting) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, for example esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts absorption and distribution of study drugs (for example, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs.
* Have a history or presence of thyroid disease.
* Show history or evidence of significant active neuropsychiatric disease.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Intend to use over-the-counter medication within 7 days prior to dosing or prescription medication (with the exception of vitamin/mineral supplements and/or hormone replacement therapy) within 14 days prior to dosing.
* Use drugs that are known substrates, inducers, or inhibitors of cytochrome P450 (CYP) enzyme pathways or phosphorylated glycoprotein (P-gp) within 14 days prior to the first dose.
* Have donated blood of more than 500 mL within the month prior to screening.
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), and are subjects unwilling to stop alcohol consumption from 48 hours before Admission (Day -1) until discharge from the unit for each treatment period, and to limit alcohol intake to a maximum of 2 units/day on all other days from screening through 48 hours prior to the post-study visit (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Are subjects who, in the opinion of the investigator, are in any way unsuitable to participate in the study.
* Are women of child bearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] de la Pena A, Cui X, Geiser J, Loghin C. No Dose Adjustment is Recommended for Digoxin, Warfarin, Atorvastatin or a Combination Oral Contraceptive When Coadministered with Dulaglutide. Clin Pharmacokinet. 2017 Nov;56(11):1415-1427. doi: 10.1007/s40262-017-0531-7. PMID 28357715

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2189265 + Atorvastatin: Period 1: Participants received a single 40-milligram (mg) oral dose of atorvastatin on Day 1, followed by a 7- to 10-day washout period between Day 1 of Period 1 and Day 1 of Period 2.
  Period 2: Participants received a single 1.5-mg subcutaneous dose of LY2189265 on Day 1, followed by a single 40-mg oral dose of atorvastatin on Day 3.
Period: Overall Study
Arm/Group | LY2189265 + Atorvastatin
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LY2189265 + Atorvastatin
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Atorvastatin: Maximum Plasma Concentration (Cmax)
Time Frame: Pre-dose to 56 hours post-dose
Population: All randomized participants who received at least 1 dose of study drug and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 40 mg Atorvastatin Alone: Period 1: Participants received a single 40-milligram (mg) oral dose of atorvastatin on Day 1, followed by a 7- to 10-day washout period between Day 1 of Period 1 and Day 1 of Period 2.
- 1.5 mg LY2189265 + 40 mg Atorvastatin: Period 2: Participants received a single 1.5-mg subcutaneous dose of LY2189265 on Day 1, followed by a single 40-mg oral dose of atorvastatin on Day 3.
Arm/Group | 40 mg Atorvastatin Alone | 1.5 mg LY2189265 + 40 mg Atorvastatin
Number analyzed (Participants) | 27 | 27
nanogram per milliliter (ng/mL) | 19.5 (60) | 5.78 (86)

2. Primary Outcome: Pharmacokinetics of Atorvastatin: Area Under the Curve (AUC)
Description: This measure is based on the pharmacokinetic area under the atorvastatin plasma concentration-time curve from time 0 to infinity.
Time Frame: Pre-dose to 56 hours post-dose
Population: All randomized participants who received at least 1 dose of study drug and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 40 mg Atorvastatin Alone | 1.5 mg LY2189265 + 40 mg Atorvastatin
Number analyzed (Participants) | 27 | 26
nanogram*hour per milliliter (ng*h/mL) | 82.8 (33) | 65.9 (35)

3. Secondary Outcome: Pharmacokinetics of Para-Hydroxyatorvastatin: Maximum Concentration (Cmax)
Time Frame: Pre-dose to 56 hours post-dose
Population: All randomized participants who received at least 1 dose of study drug and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 40 mg Atorvastatin Alone | 1.5 mg LY2189265 + 40 mg Atorvastatin
Number analyzed (Participants) | 27 | 26
nanogram per milliliter (ng/mL) | 0.473 (81) | 0.360 (69)

4. Secondary Outcome: Pharmacokinetics of Para-Hydroxyatorvastatin: Area Under the Curve (AUC)
Description: This measure is based on the pharmacokinetic area under the para-hydroxyatorvastatin concentration-time curve from time 0 to infinity. The outcome is not available for this metabolite since the terminal elimination phase was not determinable.
Time Frame: Pre-dose to 56 hours post-dose
Population: No participants were analyzed for this outcome measure since the terminal elimination phase was not determinable.
Arm/Group | 40 mg Atorvastatin Alone | 1.5 mg LY2189265 + 40 mg Atorvastatin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pharmacokinetics of Ortho-Hydroxyatorvastatin: Maximum Concentration (Cmax)
Time Frame: Pre-dose to 56 hours post-dose
Population: All randomized participants who received at least 1 dose of study drug and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 40 mg Atorvastatin Alone | 1.5 mg LY2189265 + 40 mg Atorvastatin
Number analyzed (Participants) | 27 | 27
nanogram per milliliter (ng/mL) | 14.4 (46) | 5.66 (60)

6. Secondary Outcome: Pharmacokinetics of Ortho-Hydroxyatorvastatin: Area Under the Curve (AUC)
Description: This measure is based on the pharmacokinetic area under the ortho-hydroxyatorvastatin concentration-time curve from time 0 to infinity.
Time Frame: Pre-dose to 56 hours post-dose
Population: All randomized participants who received at least 1 dose of study drug and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 40 mg Atorvastatin Alone | 1.5 mg LY2189265 + 40 mg Atorvastatin
Number analyzed (Participants) | 27 | 27
nanogram*hour per milliliter (ng*h/mL) | 102 (30) | 95.9 (28)

ADVERSE EVENTS:
Groups:
- 1.5 mg LY2189265: Period 2: Participants received a single 1.5-mg subcutaneous dose of LY2189265 on Day 1, followed by a single 40-mg oral dose of atorvastatin on Day 3. The time period for this arm was from Day 1 to predose of atorvastatin on Day 3.
- 1.5 mg LY2189265 + 40 mg Atorvastatin: Period 2: Participants received a single 1.5-mg subcutaneous dose of LY2189265 on Day 1, followed by a single 40-mg oral dose of atorvastatin on Day 3. The time period for this arm was after the atorvastatin dose on Day 3 in Period 2.
Arm/Group | 40 mg Atorvastatin Alone | 1.5 mg LY2189265 | 1.5 mg LY2189265 + 40 mg Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 8/27 | 23/27 | 16/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg Atorvastatin Alone (N=27) | 1.5 mg LY2189265 (N=27) | 1.5 mg LY2189265 + 40 mg Atorvastatin (N=27)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 9 (10) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (5)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (9) | 3 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (4)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 12 (12) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Needle track marks (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days